CLINICAL TRIAL: NCT04670445
Title: Improving Patient and Caregiver Understanding of Risks and Benefits of Immunotherapy for Advanced Cancer
Acronym: UPLIFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Conquer Cancer Foundation (Other)
Responsible Party: Principal Investigator, Laura Petrillo, M.D., Physician, Division of Palliative Care, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-410
Record Dates: First submitted 2020-12-03; First posted 2020-12-17 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Stage IV Melanoma; Advanced Lung Cancer; Stage IV Non-Small Cell Lung Cancer; Unresectable Non-Small Cell Lung Carcinoma; Unresectable Stage III Non-Small Cell Lung Cancer; Small Cell Lung Cancer Extensive Stage; Stage IV Merkel Cell Carcinoma; Stage IV Cutaneous Squamous Cell Carcinoma; Stage IV Basal Cell Carcinoma; Stage IV Breast Cancer; Stage IV Colorectal Cancer; Stage IV Gastric Cancer; Stage IV Esophageal Cancer; Stage IV Hepatocellular Cancer; Stage IV Renal Cell Carcinoma; Stage IV Bladder Cancer; Stage IV Head and Neck Squamous Cell Carcinoma; Stage IV Cervical Cancer; Stage IV Endometrial Cancer; Stage IV Mesothelioma; Immunotherapy; Immune Checkpoint Inhibitors
Keywords: Stage IV Melanoma; Advanced Lung Cancer; Stage IV Non-Small Cell Lung Cancer; Unresectable Non-Small Cell Lung Carcinoma; Unresectable Stage III Non-Small Cell Lung Cancer; Small Cell Lung Cancer Extensive Stage; Stage IV Merkel Cell Carcinoma; Stage IV Cutaneous Squamous Cell Carcinoma; Stage IV Basal Cell Carcinoma; Stage IV Breast Cancer; Stage IV Colorectal Cancer; Stage IV Gastric Cancer; Stage IV Esophageal Cancer; Stage IV Hepatocellular Cancer; Stage IV Renal Cell Carcinoma; Stage IV Bladder Cancer; Stage IV Head and Neck Squamous Cell Carcinoma; Stage IV Cervical Cancer; Stage IV Endometrial Cancer; Stage IV Mesothelioma; Immunotherapy; Immune Checkpoint Inhibitors
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Merkel Cell; Carcinoma, Basal Cell; Breast Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Liver Neoplasms; Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Squamous Cell Carcinoma of Head and Neck; Uterine Cervical Neoplasms; Endometrial Neoplasms; Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Refine Intervention and Study Procedure (Experimental): Small open pilot (n=10) to refine the intervention and study procedures.
  * The study will involve three surveys (one before first infusion, one after, and one six weeks later).
  * An educational video regarding the risks, benefits, and potential outcomes of immunotherapy treatment and reviewing an immunotherapy-focused QPL prior to ICI initiation or PDF alternative to the video
  * Question-prompt list (QPL) -list of suggested questions that participant can choose to raise with the oncology team.
  Interventions: Other: Educational Video and QPL List
- Educational Video and QPL List (Experimental): Randomized into Intervention Arm
  * The study will involve three surveys (one before first infusion, one after, and one six weeks later).
  * An educational video regarding the risks, benefits, and potential outcomes of immunotherapy treatment and reviewing an immunotherapy-focused QPL prior to ICI initiation or PDF alternative to the video
  * Question-prompt list (QPL) -list of suggested questions that participant can choose to raise with the oncology team.
  * Audio Recorded Conversation with oncologist
  Interventions: Other: Educational Video and QPL List
- Usual Care (Active Comparator): Randomized into Usual Care Arm
  * The "control" group will have three surveys (one before first infusion, one after, and one six weeks later)
  * Audio Recorded Conversation with oncologist
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Educational Video and QPL List — The intervention includes a 15-minute educational video and a 2- page list of suggested questions to review with oncology team about immunotherapy.
  Arms: Educational Video and QPL List; Refine Intervention and Study Procedure
Other: Usual Care — Surveys
  Arms: Usual Care

SUMMARY:
The purpose of this study is to refine and pilot test educational material developed to educate and support patients receiving immunotherapy for advanced cancer.

The intervention is an educational video and question prompt list (QPL) to promote communication between patients, caregivers, and the oncology team about the risks and benefits of immunotherapy.

DETAILED DESCRIPTION:
This two-part study will 1) refine and 2) pilot test an intervention to improve participant's and caregiver knowledge and increase communication with the oncology team about immunotherapy.

* The intervention involves watching a video developed to educate patients regarding the risks, benefits, and potential outcomes of immunotherapy treatment and reviewing an immunotherapy-focused QPL prior to ICI initiation.
* In Part 1 of this study, investigators will conduct a small open pilot to refine the intervention and study procedures.
* In Part 2, investigators will conduct a single-site pilot randomized controlled trial including 130 patients and their caregivers, to evaluate the feasibility of intervention delivery, and the preliminary efficacy of the intervention in improving patient and caregiver knowledge.

ELIGIBILITY:
Inclusion Criteria:

* All participants (Patients and Caregivers)-Table 1

  * Age 18 or older
  * Ability to read and respond in English
* Patient Inclusion Criteria (in addition to Table 1)

  * Receiving care in the MGH Cancer Center
  * Diagnosis of advanced (stage IV) melanoma or advanced, incurable lung cancer, including stage IV non-small cell lung cancer (NSCLC), unresectable stage III NSCLC, extensive-stage small cell lung cancer.
  * Plan to initiate immunotherapy with an ICI (pembrolizumab, nivolumab, ipilimumab, atezolizumab or combination), per clinician documentation in the electronic health record or study staff communication with clinician
* Caregiver Inclusion Criteria (in addition to Table 1)

  * Identified as "a supportive person involved in their cancer care" by a patient enrolled in the study

Exclusion criteria

* Major psychiatric condition or comorbid illness that prohibits participation in the study
* Cognitive impairment that prohibits provision of informed consent or participation in the study
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-01-23 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility - enrollment | Day 1
  Feasibility of the trial will be demonstrated if at least 70% of approached participants are enrolled
Feasibility, defined as completion of study activities | Baseline to 72 hours
  80% of participants randomized to the intervention watch the video and review the QPL.
Change in participant knowledge, using the Immunotherapy Knowledge Assessment | Baseline to 72 hours
  The primary outcome is participant knowledge, as measured by the Immunotherapy Knowledge Assessment, a 9-item survey with higher scores representing greater knowledge (minimum score = 0, maximum score =9). The investigators will compute the total knowledge score at baseline and 72 hours.
Change in participant knowledge, using the Immunotherapy Knowledge Assessment | Baseline to 6 weeks
  The primary outcome is participant knowledge, Immunotherapy Knowledge Assessment, a 9-item survey with higher scores representing greater knowledge (Minimum score = 0, maximum score = 9). The investigators will compute the total knowledge score at baseline and 6 weeks.

SECONDARY OUTCOMES:
Change in participant anxiety, using the State Subscale of the State and Trait Anxiety Inventory | Baseline to 72 hours
  The investigators will use the State Subscale of the State and Trait Anxiety Inventory and baseline and 72 hours. Higher scores indicate greater anxiety (minimum score = 20, maximum score = 80).
Change in participant anxiety, using the State Subscale of the State and Trait Anxiety Inventory | Baseline to 6 weeks
  The investigators will use the State Subscale of the State and Trait Anxiety Inventory and baseline and 6 weeks. Higher scores indicate greater anxiety (minimum score = 20, maximum score = 80)
Patient questions asked in visit with oncologist | 72 hours
  The number of questions asked by patients and caregivers will be assessed by coding the transcripts of audio-recorded oncology visits and compared between arms using the negative binomial model.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Petrillo, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation